CLINICAL TRIAL: NCT00313534
Title: A Phase I Study of NDGA in Patients With Non-Metastatic Biochemically Relapsed Prostate Cancer
Brief Title: Nordihydroguaiaretic Acid in Treating Patients With Nonmetastatic Relapsed Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Ran out of drug
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000455645; UCSF-035510; UCSF-H45860-23712-02A
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage I prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Masoprocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: masoprocol

SUMMARY:
RATIONALE: Nordihydroguaiaretic acid may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of nordihydroguaiaretic acid in treating patients with nonmetastatic relapsed prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of nordihydroguaiaretic acid (NDGA) in patients with nonmetastatic, biochemically relapsed prostate cancer.

Secondary

* Determine prostate-specific antigen-modulating effects of NDGA in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral nordihydroguaiaretic acid (NDGA) twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of NDGA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer, meeting 1 of the following criteria:

  * Androgen-dependent disease (testosterone ≥ 250 ng/mL)
  * Androgen-independent disease (testosterone < 50 ng/mL)
* Received prior definitive therapy for primary prostate cancer comprising any of the following:

  * External-beam radiotherapy with or without hormonal therapy
  * Brachytherapy with or without pelvic external-beam radiotherapy or hormonal therapy
  * Radical prostatectomy with or without adjuvant or salvage radiotherapy
  * Cryotherapy
* Must have evidence of disease progression, as evidenced by elevated prostate-specific antigen (PSA) that has risen serially from post-definitive therapy nadir on 2 determinations taken ≥ 1 week apart

  * Elevated PSA, meeting 1 of the following criteria:

    * At least 1.0 ng/mL post radiotherapy or cryotherapy
    * At least 4 ng/mL post radical prostatectomy
  * Must show disease progression after discontinuation of the antiandrogen (for patients with androgen-dependent disease receiving antiandrogen as part of primary androgen ablation)
* No metastatic disease, confirmed by negative bone scan and negative CT scan or MRI of abdomen/pelvis

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST ≤ 1.5 times ULN
* No other medical condition that would interfere with study therapy or compliance
* No other active malignancy except previously treated squamous cell or basal cell skin cancer or cancer that has been treated and considered to be at < 30% risk of relapse
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 8 weeks since prior strontium-chloride Sr 89
* More than 4 weeks since first dose of bisphosphonates
* More than 4 weeks since prior major surgery or radiotherapy
* At least 4 weeks since prior hormonal agents, including megestrol or steroids

  * Concurrent luteinizing hormone-releasing hormone analogs allowed to maintain castrate levels of testosterone
* At least 4 weeks since prior and no concurrent saw palmetto, finasteride, or any herbal agent intended to lower PSA
* Prior adjuvant or neoadjuvant androgen-deprivation therapy allowed for androgen-dependent prostate cancer provided that all of the following are met:

  * No more than 8 months of androgen deprivation
  * At least 12 months since last day of effective androgen deprivation
  * Testosterone > 250 ng/mL at enrollment
* Prior hormonal therapy, chemotherapy, or investigational therapy for biochemical relapse allowed
* No concurrent chemotherapeutic, immunotherapeutic, or other investigational agents
* No concurrent radiotherapy
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity as measured by CTC v3.0

SECONDARY OUTCOMES:
Maximum tolerated dose
Prostate-specific antigen (PSA) at baseline and on day 1 of each course

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ryan, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States